CLINICAL TRIAL: NCT04465110
Title: Effects of Chronic Dietary Grape Seed Extract Supplementation on Aortic Stiffness and Hemodynamic Responses in Obese/Overweight Males During Submaximal Exercise
Brief Title: Effects of Chronic Dietary Grape Seed Extract Supplementation on Aortic Stiffness and Hemodynamic Responses to Exercise in Obese Males
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: California Baptist University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 109-1819-EXP
Record Dates: First submitted 2020-07-06; First posted 2020-07-09 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Obesity Adult Onset
MeSH Terms: interventions — Grape Seed Extract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GSE group (Experimental): Subjects took a single dose of 600 mg GSE in capsule form through ingestion 7 days
  Interventions: Dietary Supplement: Grape Seed Extract
- Placebo group (Placebo Comparator): Subjects took a single dose of 600 mg starch in capsule form through ingestion 7 days
  Interventions: Dietary Supplement: Grape Seed Extract

INTERVENTIONS:
Dietary Supplement: Grape Seed Extract — Subjects took a single dose of 600 mg GSE in capsule form through ingestion 2 hours prior to testing Dietary Supplement: Grape seed extract Two capsule grape seed extract (total 600 mg) per day

SUMMARY:
It was demonstrated that acute dietary supplementation with GSE reduced arterial blood pressure via reduction in Q in obese individuals. However, no studies have investigated the chronic effects of dietary GSE supplementation on hemodynamic responses during exercise. Given the fact that obesity is associated with an impaired function of eNOS, the effect of chronic dietary GSE supplementation on abnormal blood pressure response to exercise and aortic stiffness (AoS) needs be elucidated. Thus, it is hypothesized that GSE decreases systolic blood pressure (SBP), diastolic blood pressure (DBP), mean arterial pressure (MAP), Q, and aortic stiffness at rest and during exercise. This study would determine that this supplementation may be used as a non-pharmacological intervention to prevent incident hypertension and cardiovascular events during exercise via enhanced endothelial function.

DETAILED DESCRIPTION:
We investigated whether elevated blood pressure and aortic stiffness (AoS) characterized in obese and overweight males (N=10) are reduced following chronic GSE supplementation during exercise. Systolic blood pressure (SBP), diastolic blood pressure (DBP), mean arterial pressure (MAP), heart rate (HR), stroke volume (SV), cardiac output (Q), total vascular conductance (TVC), and AoS to two submaximal cycling exercises (40% and 60% VO2peak) were compared 7 days after ingestion of GSE or placebo (PL) within an one week washout period. Compared with PL, GSE supplementation significantly decreased MAP at rest, 40%, and 60% workloads. AoS was significantly reduced at rest. Q tended to be decreased, but there was no significant difference. GSE had no effect on HR, TVC, and SV. Our study indicates that chronic supplementation with GSE reduces arterial pressure at rest and during exercise primarily via the combined reduction of AoS and Q. Thus, GSE can be a dietary supplement to treat augmented blood pressure responses in obese and overweight males at rest and during exercise.

ELIGIBILITY:
Inclusion Criteria:

* Overweight: 25-29.9 kg/m2
* Obese: > 30 kg/m2
* Waist circumference: > 90 cm

Exclusion Criteria:

* Antihypertensive medication
* Major systemic disease (cancer)
* Musculoskeletal diseases
* Cardiovascular diseases or symptoms including chest pain
* Myocardial infarction
* Arrhythmias
* Heart failure

Ages: 18 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-04-22 (Actual); Study Completion 2020-04-22 (Actual)

PRIMARY OUTCOMES:
change in heart rate at rest and during exercise | 7 day supplementation
  beats per minute
change in stroke volume at rest and during exercise | 7 day supplementation
  volume per stroke
change in cardiac output at rest and during exercise | 7 day supplementation
  total volume for one minute
change in systolic blood pressure at rest and during exercise | 7 day supplementation
  pressure exerted during contraction
change in diastolic blood pressure at rest and during exercise | 7 day supplementation
  pressure exerted during relaxation
change in total vascular conductance at rest and during exercise | 7 day supplementation
  one reported value (cardiac output/mean arterial pressure)
change in aortic stiffness at rest | 7 day supplementation
  Arbitrary unit

CONTACTS AND LOCATIONS:
Overall Officials: Jong-Kyung Kim, Ph.D, Principal Investigator — California Baptist University
Locations (1):
- California Baptist University, Riverside, California, United States

IPD SHARING:
Plan to Share IPD: Yes
To determine the chronic effects of dietary grape seed extraction, all data collected at rest and during exercise will be shared with other researchers in the publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: All data will be available after publication
Access Criteria: People can access the data based on the copyright of a journal after its publication.
URL: https://pubmed.ncbi.nlm.nih.gov/

REFERENCES:
- [Derived] Dillon K, Shariffi B, Gillum T, Boyer W, Sullivan S, Kim JK. Effects of chronic dietary grape seed extract supplementation on aortic stiffness and hemodynamic responses in obese/overweight males during submaximal exercise. Eur J Sport Sci. 2022 Jul;22(7):1057-1064. doi: 10.1080/17461391.2021.1923815. Epub 2021 May 20. PMID 33905304